CLINICAL TRIAL: NCT03508232
Title: Matrix Metalloproteinase Inhibition With Doxycycline to Prevent Adverse Remodeling After Acute Myocardial Infarction: A Pilot Study
Brief Title: Doxycycline to Protect Heart Muscle After Heart Attacks
Status: Recruiting | Phase: Phase 2 | Type: Interventional
Sponsor: University of Alberta (Other)
Collaborators: Royal Alexandra Hospital (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Prevention
Other Study IDs: DOXY-STEMI
Record Dates: First submitted 2018-04-16; First posted 2018-04-25 (Actual); Last update posted 2025-02-04 (Actual); Status verified 2025-02

CONDITIONS: ST Segment Elevation Myocardial Infarction; Heart Failure
MeSH Terms: conditions — ST Elevation Myocardial Infarction; Heart Failure | interventions — Doxycycline

STUDY DESIGN:
Intervention Model Description: Randomized, double-blinded, placebo-controlled study
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Masking Description: Double-blinding. Randomization will be done prior to the study and with binary encoding, for further blinding. Drug randomization (placebo or doxycycline) will be done by the Drug Development and Innovation Centre in the Faculty of Pharmacy and Pharmaceutical Sciences at the University of Alberta, with 50% allocated in the Placebo Control Group and 50% in the Doxycycline Group. The coding list will be generated and kept sealed by the PI. Patients will be randomized during recruitment, following a previously generated list with 50% of patients allocated to each group.
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- Placebo control (Placebo Comparator): Two placebo capsules upon enrollment, followed by one placebo capsule p.o. every 12 hours for 7 days
  Interventions: Drug: Doxycycline Hyclate
- Doxycycline hyclate (Experimental): Two 100mg doxycycline capsules (200 mg) p.o. upon enrollment, followed by one 100 mg capsule p.o. every 12 hours for 7 days
  Interventions: Drug: Placebo

INTERVENTIONS:
Drug: Placebo — Patients will receive placebo in a loading dose of two capsules initially followed by one capsule every 12 hours for 7 days.
  Arms: Doxycycline hyclate
Drug: Doxycycline Hyclate — Patients will receive doxycycline hyclate in a loading dose of two 100 mg capsules (200 mg total) initially followed by one 100 mg capsule every 12 hours for 7 days.
  Other Names: Doxycycline
  Arms: Placebo control

SUMMARY:
Current medical treatment allows more people to survive heart attacks than in the past. However, some of the survivors suffer heart disease and require hospitalization later on. The causes behind this heart disease (heart failure) after a heart attack are poorly understood.

Matrix metalloproteinase 2 (MMP-2) is a protein that cuts other proteins into pieces, and is activated in heart muscle when there is a heart attack. MMP-2 causes heart injury when the blood flow to the heart is restored after the attack. Blocking MMP-2 activity is a potential therapy to prevent heart injury under these circumstances. The only MMP-2 inhibiting drug currently approved for clinical use is doxycycline, specifically used to treat periodontitis (gum inflammation) and rosacea (a skin condition). At higher doses doxycycline also acts as an antibiotic for which it has been clinically used for decades.

A previous clinical study found that taking doxycycline twice a day, for one week after a heart attack improved the health of the patients' hearts. The investigators have conducted a similar study in patients that had surgery to replace blocked coronary arteries (blood vessels that feed the heart muscle). These patients took a low dose of doxycycline once a day for 2 days before surgery, on the day of the surgery, and three days after surgery. The participants in this study showed no adverse effects of using doxycycline.

The goal of this study is to see if doxycycline protects the hearts of patients that suffered a heart attack. All patients will receive standard clinical care for their condition, but in addition will take a doxycycline capsule twice a day, or a placebo capsule for 7 days, as soon as possible after being diagnosed with a heart attack. Three months later, the investigators will evaluate the patients by looking at their heart structure using magnetic resonance imaging (MRI). MRI is a powerful tool that allows doctors to see inside the body without surgery or X-ray radiation. The hearts of those patients that received doxycycline are expected to be healthier than those who received placebo.

The investigators plan to promote the use of doxycycline to protect the hearts of patients with heart attacks. If successful, doxycycline could help improve the quality of life of heart attack survivors.

DETAILED DESCRIPTION:
Background:

Matrix metalloproteinases (MMPs) are activated in myocardial ischemia, digesting key structural components in cardiac muscle in the setting of myocardial infarction and myocardial ischemia-reperfusion injury (Schulz, 2007, Annu. Rev. Pharmacol. Toxicol. 47, 211-42).

The antibiotic doxycycline is the only drug approved as an MMP inhibitor by Health Canada and the U.S. FDA for the treatment of periodontitis and rosacea at sub-antimicrobial doses.

Doxycycline decreases intracellular proteolysis, improves cardiac function, and reduces infarct size in animal models of ischemia-reperfusion injury (Cheung et al, 2002, Circulation 101:1833-39; Villarreal et al, 2003, Circulation 208:1487-92).

TIPTOP (Cerisano et al, 2014, Eur Heart J 35: 184-91) was a randomized open-label trial (110 patients) that studied the effect of 1-week doxycycline given post-percutaneous coronary intervention (PCI) in patients with anterior STEMI. Patients who received doxycycline showed improved echocardiographic indices at 6 months relative to untreated controls: left ventricular end diastolic volume index (LVEDVi) -8 mL ± 14 mL (P=0.004), left ventricular end systolic volume index (LVESVi) -6 mL ± 12 mL (P=0.02), and left ventricular ejection fraction (LVEF) +5% ± 12% (P=0.04). They also showed decreased infarct sizes (-6%, P=0.05) by single photon emission computed tomography (SPECT).

Rationale for study:

The TIPTOP pilot study showed promise for doxycycline therapy to decrease adverse ventricular remodeling post-PCI in STEMI patients. Animal models suggest that MMP activation occurs early in reperfusion (within 5 minutes) following severe ischemia, and the TIPTOP pilot showed that early treatment may result in measurable clinical benefit. However, the TIPTOP pilot was an open label study and used a low resolution approach to measure clinical outcomes.

This is a small-scale, single-centre Phase II trial with double blinding, and includes the use of magnetic resonance imaging to measure primary (LVESVi) and secondary outcomes (LVEF ad LVEDVi). The investigators anticipate beneficial effects of doxycycline, with patients showing lower levels of LVESVi and LVEDVi, increased LVEF by MRI, and reduced infarct sizes, compared to placebo at 3 months. The investigators also expect hospitalization and mortality rates due to cardiac events to be reduced in these patients.

If successful, the overarching goal is to develop a multi-center randomized, blinded, placebo-controlled trial to examine the effect of early doxycycline therapy in the setting of STEMI.

ELIGIBILITY:
Inclusion Criteria:

1. 18+ year old
2. Diagnosis of acute ST-elevation myocardial infarction (STEMI)
3. Primary STEMI
4. Symptom onset of less than 12 hours
5. Admitted to the Royal Alexandra Hospital in Edmonton, Alberta

Exclusion Criteria:

1. Low risk inferior STEMI (total ST elevation plus depression <4mm)
2. Cardiogenic shock
3. Use of thrombolytics
4. Prior history of myocardial infarction or heart failure
5. Known hypersensitivity to tetracyclines
6. Any concurrent medical condition expected to reduce life expectancy to <1 year
7. Symptom onset to treatment (loading dose) time longer than 24 hours
8. Poor renal function (eGFR<30 mL/min/1.73m2) or other contraindications to MRI (claustrophobia, pregnancy, PPM/ICD, sub-arachnoid clips, retained ocular foreign body)

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 170 (Estimated)
Dates: Start 2020-01-06 (Actual); Primary Completion 2025-12-31 (Estimated); Study Completion 2025-12-31 (Estimated)

PRIMARY OUTCOMES:
Left ventricular end-systolic volume index (LVESVi) | 3 months post intervention
  Left ventricular end-systolic volume index (LVESVi) measured by magnetic resonance imaging (MRI) at 3 months post intervention

SECONDARY OUTCOMES:
Composite endpoint of mortality and hospital admission due to re-infarction, heart failure, or stroke | 3 months and one year post intervention
  Composite endpoint of mortality and hospital admission due to re-infarction, heart failure, or stroke at 3 months and 1 year.
Left ventricular ejection fraction (LVEF) | 3 months post intervention
  Left ventricular ejection fraction (LVEF) by cardiac MRI and echocardiography during hospital admission and at 3-month follow-up.
Left ventricular end-diastolic volume index (LVEDVi) | 3 months post intervention
  Left ventricular end-diastolic volume index (LVEDVi) by cardiac MRI and echocardiography during hospital admission and at 3-month follow-up.
Infarct size | 3 months post intervention
  Infarct size by cardiac MRI during hospital admission and at 3-month follow-up

CONTACTS AND LOCATIONS:
Overall Officials: Richard Schulz, PhD, Study Chair — Dept. of Pediatrics and Pharmacology, University of Alberta; Peter Hwang, MD, PhD, Study Director — Dept. of Medicine, University of Alberta; Benjamin Tyrrell, MD, Study Director — Dept. of Medicine, University of Alberta; Richard Coulden, MD, Principal Investigator — Dept. of Radiology and Diagnostic Imaging, University of Alberta; Neil Brass, MD, Principal Investigator — Dept. of Medicine, University of Alberta; Raymond Leung, MD, Principal Investigator — CK Hui Heart Centre, Royal Alexandra Hospital, Edmonton, Alberta.; Kevin Bainey, MD, Principal Investigator — Dept. of Medicine, University of Alberta; Richard Thompson, MD, Principal Investigator — Dept. of Biomedical Engineering, University of Alberta; Ian Paterson, MD, Principal Investigator — Dept. of Medicine, University of Alberta
Locations (1):
- Royal Alexandra Hospital, Edmonton, Alberta, Canada

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Schulz R. Intracellular targets of matrix metalloproteinase-2 in cardiac disease: rationale and therapeutic approaches. Annu Rev Pharmacol Toxicol. 2007;47:211-42. doi: 10.1146/annurev.pharmtox.47.120505.105230. PMID 17129183
- [Background] Cheung PY, Sawicki G, Wozniak M, Wang W, Radomski MW, Schulz R. Matrix metalloproteinase-2 contributes to ischemia-reperfusion injury in the heart. Circulation. 2000 Apr 18;101(15):1833-9. doi: 10.1161/01.cir.101.15.1833. PMID 10769285
- [Background] Villarreal FJ, Griffin M, Omens J, Dillmann W, Nguyen J, Covell J. Early short-term treatment with doxycycline modulates postinfarction left ventricular remodeling. Circulation. 2003 Sep 23;108(12):1487-92. doi: 10.1161/01.CIR.0000089090.05757.34. Epub 2003 Sep 2. PMID 12952845
- [Background] Schulze CJ, Castro MM, Kandasamy AD, Cena J, Bryden C, Wang SH, Koshal A, Tsuyuki RT, Finegan BA, Schulz R. Doxycycline reduces cardiac matrix metalloproteinase-2 activity but does not ameliorate myocardial dysfunction during reperfusion in coronary artery bypass patients undergoing cardiopulmonary bypass. Crit Care Med. 2013 Nov;41(11):2512-20. doi: 10.1097/CCM.0b013e318292373c. PMID 23928836
- [Background] Cerisano G, Buonamici P, Valenti R, Sciagra R, Raspanti S, Santini A, Carrabba N, Dovellini EV, Romito R, Pupi A, Colonna P, Antoniucci D. Early short-term doxycycline therapy in patients with acute myocardial infarction and left ventricular dysfunction to prevent the ominous progression to adverse remodelling: the TIPTOP trial. Eur Heart J. 2014 Jan;35(3):184-91. doi: 10.1093/eurheartj/eht420. Epub 2013 Oct 8. PMID 24104875